CLINICAL TRIAL: NCT03528213
Title: Utility of Sodium Lactate Infusion During Septic Shock: Pilot Study
Brief Title: Utility of Sodium Lactate Infusion During Septic Shock
Acronym: ULIS1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_56; 2017-002393-39 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
Keywords: sepsis; fluid balance; metabolism; ischemia-reperfusion; treatment
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Sodium Lactate; Saline Solution

STUDY DESIGN:
Intervention Model Description: bolus then continuous infusion of molar sodium lactate (2 doses) or normal saline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal saline (Sham Comparator): at physician discretion
  Interventions: Drug: Normal saline
- Sodium lactate light dose (Experimental): bolus 2.5ml/kg lactate 60min then 0.25ml/kg/h during 24hrs
  Interventions: Drug: Sodium Lactate light dose
- Sodium lactate high dose (Experimental): bolus 2.5ml/kg lactate 60min then 0.50ml/kg/h during 24hrs
  Interventions: Drug: Sodium Lactate high dose

INTERVENTIONS:
Drug: Sodium Lactate light dose — bolus 2.5ml/kg then 0.25ml/kg/h
  Arms: Sodium lactate light dose
Drug: Sodium Lactate high dose — bolus 2.5ml/kg then 0.5ml/kg/h
  Arms: Sodium lactate high dose
Drug: Normal saline — normal saline at physician discretion
  Arms: Normal saline

SUMMARY:
ULIS-1 is an open-label pilot study concerning utility of molar sodium lactate in fluid balance in septic shock patients

DETAILED DESCRIPTION:
ULIS-1 consists in three arms of treatment during the first 24hrs of septic shock treatment.

* normal saline
* sodium lactate 2.5ml/kg in 60min then
* either 0.25 or 0.5ml/kg/h during 24hrs Main criteria is fluid balance at 48hrs

ELIGIBILITY:
Inclusion Criteria:

* Presence of septic shock
* requiring vascular filling within 12 hours after introduction of Noradrenaline. Septic shock is defined as sepsis with persistent hypotension requiring the administration of vasopressors to maintain RTE > 65mmHg.
* social insurance

Exclusion Criteria:

* pregnancy
* cardiac arrest
* more than 50ml/kg of fluid loading
* chronic renal failure with chronic hemodialysis or the investigators estimate a need for renal replacement therapy in the following 24hrs
* child C or acute liver failure with PT<40% (unless AVK)
* plasmatic sodium <120 or >145mmol/l
* metabolic alkalosis with pH>7.45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
fluid balance | at 48 hours
  fluid balance

SECONDARY OUTCOMES:
fluid balance at day 7 | Day 7
SOFA (Sequential Organ Failure Assessment) | Day 1, Day 2, Day 3, Day 7
death in Intensive Care Unit (ICU) | Day 90
number of patients dead | Day 28
death in hospital | Day 90
catecholamines free days | Day 28
ventilator free days | Day 28
renal replacement therapy free days | Day 28
new kidney failure | Day 28
nosocomial infections | day 90
hypernatremia | Day 2
hypokaliemia | Day 2
metabolic alkalosis | day 2
hemodynamic effects assessed by the PICCO® monitoring system | at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Favory, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - CH ARRAS, Arras
  - CH DOUAI, Douai
  - Ch Dunkerque, Dunkirk
  - CH LENS, Lens
  - Hôpital Roger Salengro, CHU, Lille
  - Hopital Victor Provo - Roubaix, Roubaix
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: Undecided